CLINICAL TRIAL: NCT04921657
Title: Genome-wide Analysis of Lipid-lowering Efficacy and Drug Level of the Two Commonly Used Statins, Simvastatin and Rosuvastatin.
Brief Title: Genome-wide Analysis of Lipid-lowering Efficacy and Drug Level of Simvastatin and Rosuvastatin
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Tomlinson, Professor, Chinese University of Hong Kong
Other Study IDs: GWAS
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Hypercholesterolemia
Keywords: Statins; Pharmacogenomics
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated with statin.: Patients with hypercholesterolemia treated with rosuvastatin 10 mg daily or simvastatin 40 mg daily.
  Interventions: Drug: Rosuvastatin 10mg

INTERVENTIONS:
Drug: Rosuvastatin 10mg
  Other Names: Simvastatin 40 mg

SUMMARY:
This study will perform a genome-wide association study (GWAS) of the lipid responses to rosuvastatin and simvastatin and plasma concentrations of these two statins in a homogeneous group of Han Chinese patients.

DETAILED DESCRIPTION:
A GWAS will be performed on about 360 Han Chinese patients with hypercholesterolaemia (which may be familial or non-familial) who have previously participated in a research project on the pharmacogenetics of statins and who have been treated with rosuvastatin and simvastatin to determine the genetic factors that may be related to the reduction in plasma low-density lipoprotein cholesterol (LDL-C) and plasma concentrations of these two statins. The lipid profiles were measured at baseline on no lipid-lowering treatment and after 4-6 week treatment of rosuvastatin 10 mg daily and after treatment with simvastatin 40 mg daily for at least 6 weeks with at least a 4-week washout period between the two treatments. Plasma concentrations of these two statins and their active metabolites about 12 hours after administration of statins have been measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS).

Genotyping for the whole-genome scan will be carried out on the Illumina OminiExpress beadchip (Illumina, San Diego, CA). The samples will be processed using the Illumina iScan platform at the Li Ka Shing Institute of Health Science, The Chinese University of Hong Kong (CUHK).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypercholesterolemia (familial or non-familial)
* Eligible for statin treatment according to local guidelines in the Hong Kong Public Hospital system.

Exclusion Criteria:

* Taking other medication which may interact with the pharmacokinetics or lipid response to statins.
* Not willing to cooperate with study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypercholesterolemia attending medical clinics in Hong Kong who were eligible for statin treatment according to local guidelines in Hong Kong and willing to give informed consent for DNA analysis.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2014-11; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Genome-wide analysis of DNA sample | DNA samples taken after 4 weeks on statin treatment.
  Presence or absence of single-nucleotide polymorphisms (SNPs) at over 700,000 points on the DNA samples will be analyzed using a whole-genome scan with the Illumina Omini Express BeadChip to identify which of these SNPs are associated with the LDL cholesterol reduction with rosuvastatin.

CONTACTS AND LOCATIONS:
Overall Officials: BRIAN TOMLINSON, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Brian Tomlinson, Hong Kong, Hong Kong